CLINICAL TRIAL: NCT04564001
Title: Multicentre, Randomized, Prospective Trial Evaluating the Efficacy and Safety of Infliximab to Tocilizumab in Refractory or Relapsing Takayasu Arteritis
Acronym: INTOReTAK
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P160909
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Takayasu Arteritis
MeSH Terms: conditions — Takayasu Arteritis | interventions — Infliximab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A ( Infliximab) (Experimental): Infliximab 5mg/kg intravenously at week 0; 2; 6; 14; 22 following prescription recommendations
  Interventions: Drug: Infliximab
- B (Tocilizumab) (Experimental): Tocilizumab : 8mg/kg intravenously at week 0; 4; 8; 12; 16; 20; 24 following prescription recommendations
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Infliximab — Patients will receive infliximab 5mg/kg intravenously at week 0; 2; 6; 14; 22 in arm A
  Arms: A ( Infliximab)
Drug: Tocilizumab — Patients will receive tocilizumab 8mg/kg intravenously at week 0; 4; 8; 12; 16; 20; 24 in arm B
  Arms: B (Tocilizumab)

SUMMARY:
Takayasu arteritis (TA) is a vasculitis of unknown origin, resulting in progressive thickening and stenosis of large and medium arteries (the aorta and its major branches, and the pulmonary arteries). First line therapy of TA consists of high dose corticosteroids (CS). Between 20 and 50% of cases respond to CS alone, with subsequent resolution of symptoms and stabilization of vascular abnormalities. Although second-line agents (methotrexate, azathioprine, mercaptopurine, mycophenolate mofetil) may result in initial remission, relapses remain common when prednisone is tapered. Thus, 50% of CS-resistant or relapsing TA patients may achieve sustained remission with the addition of methotrexate. During the last decade, biologics such as anti-tumor necrosis factor alpha (anti-TNFα) and anti-interleukin-6 (anti-IL-6) have been used as third-line treatment in refractory or relapsing TA. Almost 90% of CS-methotrexate resistant TA cases responded to infliximab, an anti-TNFα, and sustained remission was obtained in 37 to 76% of the cases. Tocilizumab, an anti-IL-6 has given similar results with 68% of sustained remission in refractory TA. Irrespective of classical cardiovascular risk factors, the systemic inflammation and CS use play a pivotal role in the occurrence of cardiovascular thrombotic events (CVEs). As CVEs overlap with TA complications it is primordial to drastically taper CS in that vasculitis. We therefore hypothesize that Infliximab or Tocilizumab can achieve a remission in more than 70% of refractory/relapsing TA cases to CS associated to a second-line agent. INTOReTAK, first randomized prospective study in TA, has an original design testing Infliximab and Tocilizumab propensity to achieve over 70% of sustained remission in refractory/relapsing TA and evaluating jointly the 2 arms. The primary objective of this study is to obtain, by arm, ≥ 70% of patients at 6 months after randomization with prednisone ≤ 0.1mg/kg per day and inactive disease (NIH score ≤ 1) during the last 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Takayasu disease according to the international criteria of the American College of Rheumatology (ACR)

  * Age at disease onset < 40 years
  * Claudication of extremities
  * Decreased brachial artery pulse (one or both arteries)
  * Blood pressure difference of >10mm Hg between the arms
  * Bruit over subclavian arteries or aorta
* Active disease according to the international criteria of the National Institute of Health (NIH)
* New onset or worsening of at least two of the following four criteria

  * Systemic features
  * Elevated erythrocyte sedimentation rate
  * Features of vascular ischemia or inflammation
  * Typical angiographic features
* Refractory/relapsing disease

  * Failure of disease to respond to daily corticosteroids therapy (1mg/kg/day for > 1month), i.e. disease still active
  * Inability to taper corticosteroids below 10mg/day within 6 months
  * Inability to discontinue corticosteroids after 1 year of treatment
  * Relapse of disease after gradual decrease of corticosteroids therapy
* Patients with one immunosuppressive agent (methotrexate, azathioprine, mercaptopurine or mycophenolate mofetil)
* Age of 18 years or older
* Weight 40 - 120 kg
* Medical follow-up in a university or general hospital in France
* Social insurance
* Willing and able to provide written informed consent
* Willing and able to comply with treatment and follow-up procedures required by the study protocol
* For female subjects of child-bearing age, a negative serum pregnancy test and no pregnancy plans within 12 months
* For subjects with reproductive potential, a willingness to use contraceptive measures adequate to prevent the subject or the subject's partner from becoming pregnant during the study. Adequate contraceptive measures include hormonal methods used for two or more cycles prior to Screening (e.g., oral contraceptive pills, contraceptive patch, or contraceptive vaginal ring), barrier methods (e.g., contraceptive sponge, diaphragm used in conjunction with contraceptive foam or jelly, or condom used in conjunction with contraceptive foam or jelly), intrauterine methods (IUD), sterilization (e.g., tubal ligation or a monogamous relationship with a vasectomized partner), and abstinence.
* Chest X-ray results (postero-anterior and lateral) within 12 weeks prior to enrollment with no evidence of active tuberculosis, active infection, or malignancy
* Tuberculosis assessment:

  * Active Tuberculosis infection treatment achieved
  * Completion of at least 3 weeks treatment for Latent Tuberculosis infection
  * Negative tuberculin skin test (TST) or interferon-gamma release assay (IGRA) (e.g., QuantiFERON®-TB Gold or T-spot TB® Test)

Exclusion Criteria:

* Active tuberculosis or untreated latent tuberculosis
* Evidence of active infection (includes chronic infection)
* Infection requiring treatment with antibiotics within 2 weeks prior to enrollment
* Infection with human immunodeficiency virus (HIV), hepatitis C, or a positive hepatitis B surface antigen.
* Pregnancy or lactation
* Inability to comply with study guidelines
* Inability to provide informed consent
* Immunosuppressant type or dose modification within 30 days prior to enrollment
* Alcohol or drug abuse, that, in the investigator's opinion, could prevent a subject from fulfilling the study requirements or that would increase the risk of study procedures
* Severe renal insufficiency (creatinine clairance <30mL/min/1,73m2)
* Hepatic dysfunction as shown by aspartate transaminase (AST) or alanine transaminase (ALT) levels >5-fold the upper limit of normal
* Heart failure ≥ stage III / IV NYHA,
* History of any malignant neoplasm except adequately treated basal or squamous cell carcinoma of the skin, or solid tumors treated with curative therapy and disease free for at least 5 years.
* History of multiple sclerosis and/or demyelinating disorder
* History of severe allergic or anaphylactic reactions to infliximab, any chimeric murine monoclonal antibody, tocilizumab, and their respective excipients or prednisone
* History of immediate hypersensitivity reaction to iodinated and gadolinium-based contrast media
* Cytopenia: Hemoglobin < 8.5 g/dL, absolute neutrophil < 1.5 G/L, Platelet count < 80 G/L
* Any live (attenuated) vaccine fewer than 4 weeks before enrolment. Recombinant or killed virus vaccines fewer than 2 weeks before enrolment.
* Use of the following systemic treatments during the specified periods

  1. Treatment with biologic therapy (infliximab, adalimumab, certolizumab pegol, golimumab, anakinra, tocilizumab, etanercept, abatacept, ixekizumab, secukinumab, ustekinumab, alemtuzumab) within 6 months prior to enrollment
  2. Past treatment with rituximab within the past 12 months, or past treatment with rituximab more than 12 months ago where the B lymphocytes count has not returned to normal at time of enrollment
  3. Treatment with any systemic alkylating agents within 6 months prior to enrollment (e.g., cyclophosphamide, chlorambucil)
* Lack of affiliation to a social security benefit plan (as a beneficiary or assignee)
* Presence of any of the following disease processes:

  * Microscopic polyangiitis
  * Granulomatosis with polyangiitis
  * Eosinophilic granulomatosis with polyangiitis
  * Polyarteritis nodosa
  * Cogan's syndrome
  * Behcet's disease
  * Sarcoidosis
  * Kawasaki's disease
  * Atypical mycobacterial infections
  * Deep fungal infections
  * Lymphoma, lymphomatoid granulomatosis, or other type of malignancy tha mimics vasculitis
  * Cryoglobulinemic vasculitis
  * Systemic lupus erythematosus
  * Rheumatoid arthritis
  * Mixed connective tissue disease or any overlap autoimmune syndrome
  * Known constitutive immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with prednisone ≤ 0.1mg/kg per day and sustained inactive disease (NIH score ≤ 1) from M3 to M6 and same biological therapy from randomization | at 6 months after randomization

SECONDARY OUTCOMES:
Incidence of relapse as defined by the NIH criteria | between 3 and 6 months
Incidence of traitement failure | at 3 months after randomization
  Traitment failure will be defined as disease still active according to the NIH criteria
Incidence of revascularization procedures | at 6 months after randomization
Incidence of revascularization procedures | at 12 months after randomization
Cumulative doses of prednisone | at 6 months after randomization
Cumulative doses of prednisone | at 12 months after randomization
Incidence of adverse events of grades III and IV | at 6 months after randomization
Incidence of adverse events of grades III and IV | at 12 months after randomization
Quality of life will be assessed using the SF36 questionnaire | at 6 months
Quality of life | at 12 months
  Quality of life will be assessed using the SF36 questionnaire
Proportion of new vascular lesions | at 6 months
Proportion of new vascular lesions | at 12 months

IPD SHARING:
Plan to Share IPD: Undecided